CLINICAL TRIAL: NCT05913765
Title: Air Filtration to Improve Indoor Air Quality (IAQ) and Chronic Obstructive Pulmonary Disease (COPD) Outcomes in a High-risk Urban Population of U.S. Military Veterans
Brief Title: Air Filtration for COPD in VA Population of Veterans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: Jesse Brown VA Medical Center (U.S. Federal Agency); US Department of Housing and Urban Development (U.S. Federal Agency); Elevate (Unknown)
Responsible Party: Principal Investigator, Brent Stephens, Professor and Department Chair, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: irb-2022-92; ILHHU0049-19 (Other Grant/Funding Number: US Department of Housing and Urban Development); IRB #1675992 (Other: JBVAMC)
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, placebo-controlled case-control design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): an air cleaner with HEPA and carbon filter installed
  Interventions: Device: Air cleaner
- Placebo (Placebo Comparator): an air cleaner with the primary filter removed
  Interventions: Device: Air cleaner

INTERVENTIONS:
Device: Air cleaner — Austin Air Healthmate air cleaner with or without standard filter

SUMMARY:
The goal of this study is to investigate the effectiveness of stand-alone air filtration for improving indoor air quality (IAQ) and chronic obstructive pulmonary disease (COPD) outcomes in a high-risk urban cohort of 80 U.S. military veterans with COPD. Secondary goals of the study are to (1) investigate housing-related factors that may contribute to COPD exacerbation, (2) investigate the utility of using low-cost sensors for indoor air pollution epidemiology studies and for providing actionable or useful information on the quality of their indoor air to patients and their physicians, and (3) evaluate the costs and benefits of using stand-alone air filtration to improve IAQ and COPD outcomes.

DETAILED DESCRIPTION:
The study will utilize a randomized, single-blind, placebo-controlled case-control design in which stand-alone portable air cleaners will be introduced to the study population over a period of approximately 1 year. One-half of the study population (40 participants) will receive a normally functioning filtration unit (i.e., an air cleaner with HEPA filter installed) and one-half of the study population (40 participants) will receive a placebo filtration unit (i.e., an air cleaner with the primary filter removed). The participants will be blinded; they will not know the status of the filter. Stand-alone portable air cleaning units containing HEPA filters and high clean air delivery rates (CADRs) sufficiently sized for the spaces they will serve will be used. The study will also involve housing condition assessments conducted in each home to characterize housing-related factors that may contribute to COPD exacerbation at baseline, as well as measurements of indoor and outdoor air quality and environmental conditions, and records of clinical outcomes (e.g., COPD exacerbations, emergency room visits, 6-minute walk distance, oxygen saturation, etc. accessed through the subject's VA medical record) throughout the study duration. The validated and extensively used St. George's Respiratory Questionnaire (SGRQ-C) and Veterans RAND 36-Item Health Survey (VR-36) will be used to determine health-related quality of life (HR-QoL) of participants by the JBVAMC Study Personnel. Clinical outcomes will also be used to assess costs of care with and without filtration interventions in this population. Low-cost air quality sensors will be used to monitor IAQ for the duration of the study). The study will also evaluate the upfront costs and operational and maintenance costs of the air cleaners over the course of the intervention periods and will compare them to the expected impacts on costs of care both with and without filtration interventions in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 90+ years.
2. English speaking and writing.
3. Able to provide consent.
4. Resident of Chicago metropolitan area.
5. Veteran receiving health care at JBVAMC with a documented diagnosis of COPD.
6. Stable housing for at least 6 months prior to screening.
7. Able to communicate regularly by telephone.

Exclusion Criteria:

1. Home palliative care.
2. Life expectancy <6 months.
3. Hazardous conditions and/or safety concerns in or around the veteran's household
4. Screened patients that already have an air cleaner and alike in his/her current residence
5. Concomitant operation of a non-study air cleaner and alike by a participant in his/her current residence at any time during the course of the trial constitutes protocol violation leading to disqualification of said participant from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbations | Through study completion, an average of 1 year
  Physician diagnosed exacerbation of acute COPD

SECONDARY OUTCOMES:
ED visits | Through study completion, an average of 1 year
  Number of emergency room visits
Urgent care visits | Through study completion, an average of 1 year
  Number of urgent care visits
Unscheduled clinic visits | Through study completion, an average of 1 year
  Number of unscheduled clinic visits
6MWD | At the end of study completion, an average of 1 year
  6-minute walk distance
O2 sat | At the end of study completion, an average of 1 year
  Transcutaneous oxygen saturation at rest and during 6MWD
Health related quality of life | At the end of study completion, an average of 1 year
  Veterans Rand 36 Item Healthy Survey (VR 36)
St. George's | At the end of study completion, an average of 1 year
  St. George's Respiratory Questionnaire (SGRQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Israel Rubinstein, MD, Principal Investigator — Jesse Brown VA Medical Center; Mohammad Heidarinejad, PhD, Principal Investigator — Illinois Institute of Technology; Zane Elfessi, PharmD, Principal Investigator — Jesse Brown VA Medical Center; Kaveeta Jagota, Study Director — Jesse Brown VA Medical Center
Locations (1):
- Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephens B, Kang I, Jagota K, Elfessi Z, Karpen N, Farhoodi S, Heidarinejad M, Rubinstein I. Study protocol for a 1-year, randomized, single-blind, parallel group trial of stand-alone indoor air filtration in the homes of US military Veterans with moderate to severe COPD in metropolitan Chicago. Trials. 2025 Jun 4;26(1):196. doi: 10.1186/s13063-025-08880-0. PMID 40468409